CLINICAL TRIAL: NCT03047291
Title: Clinical and Microbiological Evaluation of the Effect of Probiotic Lactobacillus Reuteri Prodentis in the Treatment of Mucositis and Periimplantitis
Brief Title: Effect of Probiotic Lactobacillus Reuteri in the Treatment of Mucositis and Periimplantitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, MARTA GALOFRÉ MERCADÉ, DDS, MS, Associated Professor, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Universitat Internacional
Record Dates: First submitted 2017-01-29; First posted 2017-02-08 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Mucositis; Peri-implantitis
Keywords: mucositis, periimplantitis, probiotic
MeSH Terms: conditions — Mucositis; Peri-Implantitis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: A randomized controlled, parallel design, triple-blind prospective clinical study with a follow-up of 3 months.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients, the clinical examiner, the laboratory technician and the statistician did not know the content of the containers (probiotic or placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: placebo oral tablet (Placebo Comparator): Placebo tablets. Intervention: 30 placebo tablets were given after the mechanical debridement of implants with mucositis and periimplantitis.
  Interventions: Device: Placebo Oral Tablet
- Test group: probiotic oral tablet (Experimental): Probiotic tablets (Periobalance®, Sunstar, Switzerland). Intervention: 30 probiotic tablets were given after the mechanical debridement of implants with mucositis and periimplantitis.
  Interventions: Drug: Probiotic

INTERVENTIONS:
Drug: Probiotic — 30 probiotic tablets were given after the mechanical debridement of implants with mucositis and periimplantitis.
  Arms: Test group: probiotic oral tablet
Device: Placebo Oral Tablet — 30 placebo tablets were given after the mechanical debridement of implants with mucositis and periimplantitis.
  Arms: Control group: placebo oral tablet

SUMMARY:
Evaluate clinically and microbiologically the effect of the oral probiotic Lactobacillus reuteri Prodentis (PerioBalance®, Sunstar, Switzerland) on implants with mucositis or periimplantitis, as a coadjuvant treatment of mechanical therapy.

DETAILED DESCRIPTION:
A total of 44 patients, 22 with mucositis and 22 with periimplantitis, were randomly assigned to either the control or the test group, so that 11 patients received placebo and 11 probiotic treatment. After the baseline clinical, radiological and microbiological examination, and once the study group was randomly assigned (probiotic or placebo), supragingival prophylaxis was performed in the mucositis group and subgingival mechanical therapy in the periimplantitis group. Then they get a container with 30 probiotic or placebo tablets and instructions on how and when to take them. At 30 and 90 days after beginning the treatment, a clinical, radiological and microbiological examination was performed.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with general good health,
* non-smokers,
* history of mild or moderate chronic periodontitis
* at least one dental implant with probing pocket depth ≥4mm together with bleeding on probing and/or suppuration, and a fixed prosthetic restoration in function for at least 12 months,
* compliance with the periodontal maintenance program,
* accessibility during all the study period and receptiveness and ability to fulfill with the protocol.

Exclusion Criteria:

* pregnant or lactating women,
* patients who required prophylaxis of bacterial endocarditis or had taken local or systemic antibiotic, anti-inflammatory, antiseptic or probiotic therapy in the previous 3 months,
* subjects who had received surgical periodontal treatment in the last 6 months,
* uncontrolled periodontal disease,
* previous or current history of alcoholism or smoking,
* treatment with bisphosphonates, neurologic deficiencies, systemic diseases such as immunodeficiencies or uncontrolled diabetes, rheumatoid, hepatic, renal, cardiovascular or infectious pathologies, radiotherapy, chemotherapy, use of any medication which can affect at periodontal level,
* lack of patient cooperation (failure to follow the treatment instructions and/or failure to attend visits),
* implants with mobility and/or radiographic bone loss ≥ 5mm and/or ≥ 50% of implant length.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-01-01; Primary Completion 2017-03-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth | Differences between baseline and 30 and 90 days will be calculated.
  The probing pocket depth was recorded, in millimeters and at six points per tooth and implant, as the distance from the gingival margin to the bottom of the periodontal pocket and peri-implant mucosa. Measurements will be performed by a masked and calibrated investigator.

SECONDARY OUTCOMES:
Plaque index | Differences between baseline and 30 and 90 days will be calculated.
  The general plaque index (PI) was recorded according to O'Leary et al., dichotomously assigning the presence or absence of plaque on four surfaces per tooth and implant. The implant plaque index (IPI) was recorded by assigning a dichotomous value to the presence or absence of plaque (1 indicating presence of plaque and 0 absence of plaque) of the implant under study. Measurements will be performed by a masked and calibrated investigator.
Bleeding on probing | Differences between baseline and 30 and 90 days will be calculated.
  The general bleeding on probing (BOP) was determined according to Ainamo and Bay, evaluating dichotomously the presence or absence of bleeding on the mesial, distal, buccal and lingual/palatal dental or implant surfaces. The implant bleeding on probing (BOPI) was recorded using a dichotomous value depending on whether the implant under study presented bleeding or not (1 indicated bleeding and 0 no bleeding). Measurements will be performed by a masked and calibrated investigator.
Microbiological tests | Differences between baseline and 30 and 90 days will be calculated.
  Microbiological tests were performed in the deepest periimplant pocket, using the Guidor Perio-Implant Diagnostic Test® (Sunstar S.A, Switzerland), which by means of Real-Time PCR identified and quantified the total bacterial load of A. actinomycetemcomitans (DSM 8324), T. forsythia (CIP 105220), P. gingivalis (DSM 20709), T. denticola (DSM 14222), P. intermedia (DSM 20706), P. micros (DSM 20468), F. nucleatum (DSM 20482), C. rectus (LMG 18530) and E. corrodens (DSM 8340). Measurements will be performed by a masked and calibrated investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Galofré Mercadé, Principal Investigator — Universitat Internacional de Catalunya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vivekananda MR, Vandana KL, Bhat KG. Effect of the probiotic Lactobacilli reuteri (Prodentis) in the management of periodontal disease: a preliminary randomized clinical trial. J Oral Microbiol. 2010 Nov 2;2. doi: 10.3402/jom.v2i0.5344. PMID 21523225
- [Background] Flichy-Fernandez AJ, Ata-Ali J, Alegre-Domingo T, Candel-Marti E, Ata-Ali F, Palacio JR, Penarrocha-Diago M. The effect of orally administered probiotic Lactobacillus reuteri-containing tablets in peri-implant mucositis: a double-blind randomized controlled trial. J Periodontal Res. 2015 Dec;50(6):775-85. doi: 10.1111/jre.12264. Epub 2015 Feb 25. PMID 25712760
- [Background] Hallstrom H, Lindgren S, Widen C, Renvert S, Twetman S. Probiotic supplements and debridement of peri-implant mucositis: a randomized controlled trial. Acta Odontol Scand. 2016;74(1):60-6. doi: 10.3109/00016357.2015.1040065. Epub 2015 May 8. PMID 25953193
- [Result] Vicario M, Santos A, Violant D, Nart J, Giner L. Clinical changes in periodontal subjects with the probiotic Lactobacillus reuteri Prodentis: a preliminary randomized clinical trial. Acta Odontol Scand. 2013 May-Jul;71(3-4):813-9. doi: 10.3109/00016357.2012.734404. Epub 2012 Nov 26. PMID 23176716